CLINICAL TRIAL: NCT03936920
Title: Intra and Inter Reliability and Validity of the Turkish Version of Ottowa Sitting Scale in Intensive Care Unit Survivors
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Busra Aktas, physiotherapist, Izmir Katip Celebi University
Other Study IDs: IzmırIKCU
Record Dates: First submitted 2019-04-30; First posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Intensive Care (ICU) Myopathy; Functional Disturbance
MeSH Terms: conditions — Muscular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction-Objective: Balance evaluation is one of the most important components of physical examination. Studies on equilibrium assessment in different research groups; It includes measurements that assess the seating balance, which does not require complex measurements or ambulation.

In the literature, there is no clear information about balance effect in intensive care patients who can not be ambulated due to loss of advanced muscle strength, especially in the early period.

Ottowa Sitting Scale is a scale in which the balance is evaluated in the sitting position and it has no validity and reliability in Turkish.

Therefore, the aim of this study is to examine the reliability and validity of the Ottowa Sitting Scale Turkish version between measurements and measurements.

DETAILED DESCRIPTION:
In recent years, the mortality rate has decreased in an intensive care unit with the medical and technological developments related to intensive care treatments and the rate of discharge from intensive care unit (ICU) has increased. However, as the length of hospitalization in the intensive care unit prolonged, the functionalities of the patients were restricted due to changes in the musculoskeletal and cardiovascular system. Inactivity, inflammation, the use of pharmacological agents and the presence of neuromuscular syndromes associated with the critical disease lead to decreased muscle dysfunction and exercise tolerance in patients in the intensive care unit. These changes cause the health-related quality of life to be worse in people with critical illness a few months after discharge. Balance; muscle strength is affected by changes in sensory information, postural control and vestibular arrangements from the lower extremity. Studies on equilibrium assessment in different research groups; It includes measurements that assess the seating balance, which does not require complex measurements or ambulation. In the literature, there is no clear information about balance effect in intensive care patients who can not be ambulated due to loss of advanced muscle strength, especially in the early period. The Ottowa Sitting Scale is a scale in which the balance is evaluated in the sitting position and there is no validity and reliability in Turkish. For this reason, the aim of this study is to examine the reliability and validity between measurements and measurements of the Ottowa Sitting Scale's Turkish version. More than one physiotherapist scores patients for validity between the measurements. For the validity of the measurements, a physiotherapist scores the patient twice in two weeks intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in the study
2. To understand Turkish commands
3. To be able to be independent in the previous functional status
4. Sleep at least 24 hours in intensive care

Exclusion Criteria:

1. Do not want to participate in the study
2. Central or peripheral neurological damage
3. Don't understand Turkish commands
4. Unconsciousness
5. Arrhythmia
6. Acute myocardial infarction
7. Hemodynamic instability (Blood pressure> 200 or <80; Heart rate <40 or> 130, O2 saturation <88%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 80
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Ottowa Sitting Scale | 1 day
  It is a scale that does not require ambulation, is able to maintain static sitting position in the sitting position, can move in short distance, can move long distance, body rotation ability and ability to move on the hip can be fulfilled. The scoring of each unit varies between 0-4 and the maximum score is 40.
Functional Independence Scale (FIM) | 1 day
  FIM shows the degree of independence in the basic physical and cognitive activities of the individual in daily life. FIM consists of 18 questions and mainly measures 2 parameters (1- physical / motor function, 2- cognitive / cognitive function). Each item is scored at 7 levels (1-7), 'level 1 yardım means full help, and Her level 7 lan means full independence. FIM total score is between 18-126 points. The higher the individual's score, the higher the level of independence.
Berg Balance Test | 1 day
  It consists of 14 questions in which it is evaluated whether or not the balance related tasks can be fulfilled in the changing spectrum from sitting position to standing up to one foot. 0: cannot do 4: is scored as doing independently. The total score is 56. The risk of a fall from 0 to 20 is high, the risk of a fall from 21 to 40 is considered to be low and the risk of a fall from 41 to 56 is considered low.

CONTACTS AND LOCATIONS:
Overall Officials: Ilknur Gursan, Study Director — Izmir Katip Celebi University
Locations (1):
- Izmir University of Health Sciences Dr. Suat Seren Chest Diseases and Surgery Training and Research Hospital, Izmir, Cigli, Turkey (Türkiye)